CLINICAL TRIAL: NCT04753723
Title: The Use of a Platform Wound Device for Reducing Infection in Torso and Extremity Wounds: An Interventional Clinical Trial
Brief Title: The Use of a Platform Wound Device for Reducing Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Metis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PWD-1
Record Dates: First submitted 2021-02-08; First posted 2021-02-15 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Wounds and Injury; Burn Wound; Infection Wound
MeSH Terms: conditions — Wounds and Injuries; Burns; Wound Infection | interventions — Gentamicins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Platform wound device with antibiotic (Experimental): Antibiotic cream will be applied to study wounds and then dressed with the platform wound device.
  Interventions: Combination Product: Gentamycin with Platform Wound Device
- Standard of Care (No Intervention): Study wounds will be treated per the standard of care.

INTERVENTIONS:
Combination Product: Gentamycin with Platform Wound Device — Treatment of wounds with gentamycin and covered with platform wound device.
  Arms: Platform wound device with antibiotic

SUMMARY:
This study will evaluate the safety and efficacy of a novel Platform Wound Device (PWD) in its delivery of a local antibiotic, 0.1% Gentamycin cream, to prevent or treat infection in torso and extremity wounds. The hypothesis is that the PWD will be a safe and effective method to provide topical antibiotics to a torso or extremity wound, non-inferior to the current standard of care. This treatment will reduce or rapidly eradicate infection.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled clinical trial comparing the use of a platform wound device as compared to standard of care to prevent or eliminate infection in torso and extremity wounds. Patients 18-85 years of age admitted for treatment of open wound(s) will be screened for inclusion criteria and asked to consent to participate in the randomized study. The first 10 patients will be treated with the PWD + gentamicin and will serve as a safety subset. Baseline measurement of serum antibiotic concentraion will be taken prior to PWD placement and one day after. Following the safety subset, 50 patients will be randomized to standard of care or to a single application of the PWD + gentamicin. Baseline assessments will be completed on day 0, including screening, pre-procedure wound evaluation, imaging, assessments, and specimen collection. Follow-up assessments will be completed and data gathered at days 1,2,3 and 4. All data collected of the study participants will be used to evaluate the PWD delivery of antibiotic.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater or equal to 18 and age less than or equal to 85
2. Open wound up to 500cm2 in area with evidence of infection
3. Exposure of deep dermis, subcutaneous tissue, muscle, fascia, tendon, or bone

Exclusion Criteria:

1. Pregnancy
2. Prisoner
3. Active malignancy, steroid use, or immunosuppressive therapy
4. Open fracture intimately involved with wound
5. Underlying osteomyelitis
6. Hardware or prosthetic exposure within wound
7. Exposure of major named vessels or nerves
8. Known allergy to gentamicin or other aminoglycosides

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Feasibility of treatment | 48 to 96 hours
  Demonstration of the ability to enroll patients at a single institution to either the control group, receiving standard of care, or the treatment group, receiving PWD delivery and 1 dose of antibiotic (0.1% gentamicin cream) over 48 to 96 hours.
Tolerability of treatment | 48 to 96 hours
  To demonstrate that patients are able to tolerate application of the PWD with 0.1% gentamicin cream application. Tolerability will be assessed by documentation of adverse events.

SECONDARY OUTCOMES:
Effectiveness of wound swabs | 48 to 96 hours
  To demonstrate that wound swabs are an accurate and reliable measurement of infection based on semi-quantitative wound culture results.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Baptist Medical Center, San Antonio, Texas
  - North East Baptist Hospital, San Antonio, Texas
  - Mission Trail Baptist Hospital, San Antonio, Texas
  - North Central Baptist Hospital, San Antonio, Texas